CLINICAL TRIAL: NCT06268691
Title: Control of Aedes Breeding Sites With a Dual-action Insecticidal Coating is Effective in Reducing Dengue Transmission: Cluster-randomised Controlled Trial Study
Brief Title: Sustainable Reduction of Dengue in Colombia: Vector Breeding Site Intervention With an Insecticidal Coating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rocio Cardenas Sanchez (Other)
Collaborators: Göteborg University (Other); Instituto Nacional de Salud, Colombia (Other Government); Instituto Departamental de Salud de Norte de Santander (Unknown); Universidad Francisco de Paula de Santander (Unknown)
Responsible Party: Sponsor-Investigator, Rocio Cardenas Sanchez, Researcher, University of Freiburg
Organization: University of Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ProjectCOLOMBIA-ZMG.U-Freiburg
Record Dates: First submitted 2024-01-26; First posted 2024-02-20 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Dengue; Vector Borne Diseases; Arbovirus Infections; Zika; Chikungunya Fever
Keywords: novel microencapsulated formulation; insecticides
MeSH Terms: conditions — Dengue; Vector Borne Diseases; Arbovirus Infections; Zika Virus Infection; Chikungunya Fever

STUDY DESIGN:
Intervention Model Description: A cluster randomised trial for the application of a new vector control tool (insecticide coating of water containers) was conducted in the metropolitan area of Cúcuta, Colombia. Each cluster comprising approximately 2,000 dwellings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): The study was conducted in 20 clusters of 2000 dwellings each, where 10 clusters were randomly assigned to the control arm and 10 clusters to the intervention arm
- Intervention arm (Experimental): The study was conducted in 20 clusters of 2000 dwellings each, where 10 clusters were randomly assigned to the control arm and 10 clusters to the intervention arm
  Interventions: Other: Insecticide Coating INESFLY

INTERVENTIONS:
Other: Insecticide Coating INESFLY — The IC is an aqueous solution containing polymeric microcapsules of insecticides and insect growth regulators (pyriproxyfen-PPF (0.063%) and alphacypermertrin-ACM (0.7%) in suspension, without interaction between them, developing by INESFLY Corporation, key achievement of the year 2017 TDR-WHO.
  Other Names: Coating of microencapsulated insecticides
  Arms: Intervention arm

SUMMARY:
Effective control of Aedes aegypti mosquitoes in breeding sites with high reproductive rates could have a major impact on reducing arbovirosis in endemic communities. The application of a safe, effective, low cost and sustained insecticide coating (IC) could be an affordable response to dengue for local health services. Therefore, a cluster randomised trial for the application of a new vector control tool (insecticidal coating of water containers) was conducted in the metropolitan area of Cúcuta, Colombia. The IC is an aqueous solution containing polymeric microcapsules of insecticides and insect growth regulators (pyriproxyfen-PPF (0.063%) and alphacypermertrin-ACM (0.7%) in suspension, without interaction between them, development by INESFLY®, Spain.

The main questions it aims to answer are:

Whether the control of the main breeding sites of Aedes mosquitoes, through the application of insecticide coating, in clusters of dwellings, could reduce dengue transmission in a sustainable way, compared to untreated clusters, in Cúcuta, Colombia.

Whether the control of the main breeding sites of Aedes mosquitoes through the application of insecticide coating, in clusters of dwellings, could reduce the Aedes Indices in a sustainable way, compared to untreated clusters. The initial preparation phases: i) socialization ii) A safety evaluation to determine the health risks of IC in domestic water containers; iii) The determination of the effects and efficacy of IC on Aedes aegypti.

The Baseline study to characterise the study clusters from entomological, epidemiological and socio-economic approaches was carried out in 2019-2020. The IC application phase in the intervention arm was carried out between Nov-2021 and Jan-2022, with the respective monitoring of the safety of IC use. This was followed by entomological monitoring. Finally, the 9-month post-intervention evaluation. Epidemiological data were obtained from the National Public Health Surveillance System - SIVIGILA.

The study was conducted in 20 clusters of 2000 dwellings each, where 10 clusters were randomly assigned to the control arm and 10 clusters to the intervention arm.

In order to determine the effect of IC application in household tanks, the dengue incidence and entomological indices are compared in the study clusters. The data are analysed under the difference in difference approach. Additionally, the acceptance of IC in the intervened communities and local health services is determined.

DETAILED DESCRIPTION:
1. Introduction. Arboviral diseases such as dengue, Zika and chikungunya (DZC) - transmitted by Aedes mosquitoes - are spreading rapidly around the world. Without mass availability of vaccines or specific treatments, vector control strategies are crucial to reduce transmission and prevent such diseases. Unfortunately, insecticide resistance, the high cost of control alternatives using modern technology and low community participation are major challenges for health programs. There is an urgent need to develop new effective, acceptable and sustainable interventions to reduce the incidence of DZC. In alliance with the Center for Medicine and Society in Freiburg, Germany ("Zentrum für Medizin und Gesellschaft" -ZMG) and Institute of Public Health, Gothenburg University, researchers from the National Institute of Health together with the Vector Control Group of the State Institute of Health (IDS) and GIGA group of UFPS have applied and validated in water containers, a novel vector control method called "insecticide coating (IC)" developed by researchers from the Spanish company INESFLY, under the framework of a research project that seeks to combat Aedes mosquitoes in the metropolitan area of Cúcuta, Colombia. The IC is an aqueous solution containing polymeric microcapsules of insecticides and insect growth regulators (pyriproxyfen-PPF (0.063%) and alphacypermertrin-ACM (0.7%) in suspension, without interaction between them. Its technology allows a gradual release, thus achieving less harmful products, with a high residual effect and high persistence, which makes it effective for the control of larvae and adult mosquitoes.
2. Place of study. The study was conducted in Metropolitan Cucuta in the North-East of Colombia, including the city of Cucuta (629,414), and two adjacent municipalities Villa del Rosario (93,735) and Los Patios (81,411 inhabitants) located in the Norte de Santander state.
3. This study consists of five phases. 3.1. The first phase consisted of preliminary activities, which included socializations with Colombian health managers, project referents and community leaders. A safety evaluation was carried out at one workstation by studying the leaching of alphacypermethrin and pyriproxyfen in tanks of various surfaces treated with the IC product (plastic, metal, cement-tile). In this evaluation, the dose additivity model was applied (samples were processed at the Liverpool School of Tropical Medicine, UK by Dr. Mark Paine's laboratory).

   3.2. The second phase was the experimental evaluation of the insecticidal effect of the IC on Aedes, under laboratory and semi-field conditions developed by the Entomology Group of the National Health Institute and the Entomology Unit of the State Health Institute (IDS) of Norte de Santander. Bioassays were designed to determine the following effects of IC on Aedes states: Lethal effect and sterilising effect on gravid females; Effect on egg hatching and adult emergence inhibition; Residual effect for 12 months.

   3.3. The third phase was the baseline study to collect information on the characteristics of the population, perceptions of these diseases, willingness to apply the insecticide coating in their water containers, the epidemiological profile and entomological indices (larvae and pupae/person). The sample size was calculated for detection of a 50% reduction in the House Index with > 99% power at 5% significance level. Given a baseline HI of 30%, an intra-cluster correlation coefficient (ICC) of 0.01 and a cluster size of 2,000 households it was found that a minimum of 12 clusters per study arm was needed. The same result but with a lower power (68%) was found for a baseline DZC incidence of 3% and a 50% reduction in the intervention arm. A large number of households per cluster was needed as Ae. aegypti vectors are day-biters and it was assumed that many household members stay within their neighbourhoods during the day (mainly housewives, small children and school children when the school is close to their house) where they are at risk to get infected. All estimations were done through The Shiny CRT Calculator, a web-based app to determine sample size and power for cluster trials.

   3.3.1. Sampling procedure for household survey and entomological inspections. By this way, 24 high and medium endemic areas (clusters) were selected in Cucuta (16 clusters), Los Patios (4 clusters) and Villa del Rosario (4 clusters). For the baseline study they were not yet paired and allocated to the intervention and control arm as this was planned to do with the information resulting from the baseline study enabling us to find pairs of clusters with similar characteristics (endemicity, socio-economic conditions and characteristics of public spaces) For the entomological/socio-demographic household survey, a proportion of 10% of 2000 houses was sampled in this study, resulting in 200 houses in each cluster. This number was rounded to 250 by convenience. Therefore, the study targeted 6000 households (250 households in each cluster) using a systematic random sampling method. For this we first estimated the sampling interval by dividing the total number of households in each cluster (around 2000) by the number of sample households (250), resulting in a sampling interval of 8. All households located within each cluster were mapped and a randomly defined starting point was selected and from there every 8th household was visited. 3.3.2. Data collection. The baseline surveys included a household questionnaire and entomological survey. The instruments were discussed in a participatory workshop with experts and pre-tested among the members of vector control staff in the three municipalities leading to some modifications. An extensive training was conducted by the research team before starting the field work.

   3.3.3. Household questionnaire. Demographic and health data was collected through face-to-face interviews using a standard questionnaire that included both structured and semi- structured questions. Household questionnaire was adapted from published research in Colombia. The questions referred to socio-demographic parameters (number of people living in the house, age, sex, and educational level), self-reported DZC disease acquired during the last months, population mobility during the day, usage of water in tanks and willingness to accept the intervention trial.

   3.3.4. Entomological survey. The standard entomological survey form was adapted following the guidelines of Standard Operational Procedures (SOPs) by WHO. The questions were adapted to local conditions and survey requirements. The following data were recorded from each household: total number of containers (potential breeding sites), number of mosquito larvae positive and negative containers (any species), pupae count per container, container type, and other container characteristics (if they were covered or uncovered, outdoors or indoors).

   3.3.5. Dengue surveillance and case definition. Data of the national surveillance system were obtained from SIVIGILA (the national health surveillance system), aggregated by year and setting (study areas) over the study period. This study used annual population data (from the National Institute of Statistics-DANE, for calculating the incidence rate.

   3.4. The fourth phase: intervention, monitoring and evaluation. The global information allowed the conformation of 24 clusters with 1500-2000 houses each; from which 20 clusters were selected as appropriate for the next phase.

   3.4.1. Intervention. The assignment of clusters to intervention or control status was randomized (using computer generated random numbers). The large intervention trial where the IC was applied to water containers, particularly wash tanks, targeting 20,000 households from the 10 randomly selected clusters. The other 10 control clusters do not receive the IC but received routine vector surveillance activities. 3.4.2. Monitoring. During the 12 -months observation period new cases of the 3 target diseases were monitored through the national surveillance system SIVIGILA. Vector densities through larval and pupal surveys (Pupae per Person Index) were determined in a subsample of 40 houses in each cluster (800 houses in total) at months 3 and 6.

   3.4.3. Evaluation. Nine months after the intervention, an entomological and socio-demographic survey was conducted again using the same questionnaires and methodology as in the baseline study.

   3.5. The fifth phase Data management and analysis. To base-line descriptive analyse and double data entry was practiced (to minimize data entry errors) into a database using Microsoft Office Excel software by an assistant and supervised by the research team. The analysis was done using SPSS software version 28.0.1.1. Socio-demographic data were entered into a database. We assessed the frequency of variables potentially associated with the outcomes of recent dengue virus infection (sex, age, educational level, people's mobility) and self-reported dengue fever in household members. Persons' Chi-square test (χ2) was applied to determine the differences between population characteristics and DZC self-reported cases, and peoples' mobility across all settings. All statistical analyses were performed at a 0.05 significance level. Entomological indices were analysed per cluster and overall to show the presence, distribution and abundance of Ae. aegypti and the breeding sites most productive for adult mosquitoes were identified. House index (HI): Percentage of houses infested with larvae and/or pupae. Container index (CI): Percentage of water-holding containers infested with larvae or pupae. Breteau index (BI): Number of positive containers per 100 houses inspected. Pupae per person (PPI): Number of pupae per person in each household. To estimate the pupal count for large containers (more than 20 L) the methodology by Romero-Vivas was used: According to water level, the number of pupae found was multiplied by a calibration factor. In the evaluation analysis, Difference-in-differences (DiD) approaches are applied to comparing areas before-after the intervention and between control and treatment clusters, taking into account the clustering effect, and estimating the statistical significance through the P-value. Likewise, the Reduction of dengue cases reported by SIVIGILA was estimated, according to the incidence of dengue, determining its significance and probability of certainty.
4. Ethical considerations. The household questionnaire was only applied to adults who provided information related to the purpose of this study. No child or adolescent below the age of 18 was interviewed in this study. All people participating in the study were informed in local language through the study information sheet in a written and oral way. They were asked to sign the informed consent form. All participants were informed that their participation was voluntary and that their responses remained anonymous, therefore the study used numbers which replaced the names of individuals and codes which replaced the address of the house. Before examining the domestic and peri-domestic water holding containers, the field team requested permission to enter the house, did the inspection and collected entomological and sociodemographic data. The study received approval from local health authorities in Cucuta and Norte de Santander and the study protocol was approved by the ethical committee of the Albert-Ludwigs-Universität (application number 141/19) in Freiburg, Germany and the CEMIN of National Institute of Health in Bogota, Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Dwellings located within the intervention arm
* Dwellings are inhabited
* Dwellings have a washing-tank

Exclusion Criteria:

* Dwellings that do not have washing-tanks
* Dwellings have a water tank with biological control -fish-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35000 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change of dengue incidence for 12 months | 12 months
  the dengue incidence for the year 2021 is compared with the incidence for the year 2022 in the study clusters, according to the control or intervention condition. Epidemiological data were obtained from the National Public Health Surveillance System - SIVIGILA, Norte de Santander, Colombia

SECONDARY OUTCOMES:
Change of vector densities estimated through larval and pupal indices. | 9 months
  Baseline Aedes indices are compared with post-intervention rates at 3, 6 and 9 months, and according to whether they were control or intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Kroeger, Prof. Dr., Study Director — University of Freiburg, Centre for Medicine and Society; Rocio Cardenas, Research Dr., Principal Investigator — University of Freiburg, Centre for Medicine and Society; Winfried Kern, Prof. Dr., Study Chair — University of Freiburg; Max Petzold, Prof. Dr., Study Chair — Institute of Public Health, Gothenburg University, Göteborg, Sweden
Locations (2):
- Instituto Departamental de Salud de Norte de Santander, Cúcuta, Norte de Santander Department, Colombia
- Centre for Medicine and Society, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD related to cluster results will be partially shared in the publications resulting from the study. Data may be requested with justification from the ZMG UNI-FRIEBURG researchers- data committee. Partially available at https://doi.org/10.1186/s12889-023-15893-4
Supporting Information: Study Protocol, SAP
Time Frame: up to 12 months after publication.
Access Criteria: the unit of the study is the dwelling, therefore data surveyed in dwellings, without individual addresses, will be available as supplementary material within the publications. Further data may be requested from the corresponding author up to 12 months after publication.

REFERENCES:
- [Result] Carrillo MA, Cardenas R, Yanez J, Petzold M, Kroeger A. Risk of dengue, Zika, and chikungunya transmission in the metropolitan area of Cucuta, Colombia: cross-sectional analysis, baseline for a cluster-randomised controlled trial of a novel vector tool for water containers. BMC Public Health. 2023 May 30;23(1):1000. doi: 10.1186/s12889-023-15893-4. PMID 37254133
- [Result] Carrillo MA, Kroeger A, Cardenas Sanchez R, Diaz Monsalve S, Runge-Ranzinger S. The use of mobile phones for the prevention and control of arboviral diseases: a scoping review. BMC Public Health. 2021 Jan 9;21(1):110. doi: 10.1186/s12889-020-10126-4. PMID 33422034
- [Result] Cardenas R, Hussain-Alkhateeb L, Benitez-Valladares D, Sanchez-Tejeda G, Kroeger A. The Early Warning and Response System (EWARS-TDR) for dengue outbreaks: can it also be applied to chikungunya and Zika outbreak warning? BMC Infect Dis. 2022 Mar 7;22(1):235. doi: 10.1186/s12879-022-07197-6. PMID 35255839
- [Result] Wright E, Carrillo MA, Matamoros D, Sanchez RC, Yanez J, Di Lorenzo G, Villa JM, Kroeger A. Applicability of the Mexican ovitrap system for Aedes vector surveillance in Colombia. Pathog Glob Health. 2023 Sep;117(6):554-564. doi: 10.1080/20477724.2022.2146049. Epub 2022 Nov 16. PMID 36384430
- [Result] Hussain-Alkhateeb L, Rivera Ramirez T, Kroeger A, Gozzer E, Runge-Ranzinger S. Early warning systems (EWSs) for chikungunya, dengue, malaria, yellow fever, and Zika outbreaks: What is the evidence? A scoping review. PLoS Negl Trop Dis. 2021 Sep 16;15(9):e0009686. doi: 10.1371/journal.pntd.0009686. eCollection 2021 Sep. PMID 34529649

DOCUMENTS (2):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT06268691/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT06268691/SAP_001.pdf